CLINICAL TRIAL: NCT06168149
Title: Preterm Eylem Olgularında; Fetal Akciğer Elastografi Değerlerinin Respiratuvar Distres Gelişimi Ile İlişkisi
Brief Title: The Relationship of Fetal Lung Elastography Values With the Development of Respiratory Distress in Cases of Preterm Labor
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Ahmet Kurt, Resident Physician- Obstetric and Gynecology Department, Ankara Etlik City Hospital
Other Study IDs: AEŞH-EK1-2023-516
Record Dates: First submitted 2023-11-17; First posted 2023-12-13 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Preterm Labor; Respiratory Distress Syndrome
Keywords: Preterm Labor; Respiratory Distress Syndrome; Fetal Lung Elastography; Elastography
MeSH Terms: conditions — Obstetric Labor, Premature; Respiratory Distress Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neonates with respiratory distress syndrome: A total of 80 patients with no systemic maternal disease findings and diagnoses, without chronic drug use, who were measured at least 24 hours after antenatal corticosteroids were administered during pregnancy, and whose delivery occurred within a maximum of 72 hours, will be included in our study as two case groups with and without RDS diagnosis in neonatal follow-up.
  Interventions: Diagnostic Test: fetal lung elastography measurement
- Neonates who do not develop respiratory distress syndrome: A total of 80 patients with no systemic maternal disease findings and diagnoses, without chronic drug use, who were measured at least 24 hours after antenatal corticosteroids were administered during pregnancy, and whose delivery occurred within a maximum of 72 hours, will be included in our study as two case groups with and without RDS diagnosis in neonatal follow-up.
  Interventions: Diagnostic Test: fetal lung elastography measurement

INTERVENTIONS:
Diagnostic Test: fetal lung elastography measurement — Elastography measurements are planned to be performed as in the studies "Feasibility of two-dimensional ultrasound shear wave elastography of human fetal lungs and liver: A pilot study" and "Feasibility of 2-D ultrasound shear wave elastography of fetal lungs in case of threatened preterm labour: a study protocol" in the literature examples section of the file.

SUMMARY:
The aim of this study was to compare fetal lung elastography (FAE) values between groups with and without Respiratory Distress Syndrome (RDS) in preterm neonates and to evaluate the potential of FAE to predict the risk of developing RDS.

DETAILED DESCRIPTION:
The evaluate the potential of fetal lung elastography as a non-invasive method to predict and treatment respiratory complications in preterm neonates. FAE is an imaging method that measures the elasticity properties of fetal lung tissue using ultrasound technology. This method can be helpful in providing information about the development and respiratory function of the fetal lungs.

The advantages of FAE are:

It is a non-invasive method: FAE is performed using ultrasound technology and has no known maternal or fetal harm. It stands as a potentially safe method compared to current invasive tests.

It is cost-effective and easy to perform: FAE is a procedure performed using existing ultrasound equipment at no separate cost. Therefore, it can be easily implemented and repeated in clinical settings.

Fast results: FAE provides fast results by acquiring images in real time. This indicates that FAE can be a valuable diagnostic tool in emergency situations or when rapid decision-making is required.

A potential predictive tool: The results of this study may indicate that FAE values are a potential tool for predicting the risk of developing RDS. This could be an important step to develop early diagnosis and treatment strategies to improve the respiratory health of preterm newborns.

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Single pregnant women who were followed up with a diagnosis of preterm labor between 24-33 weeks and who volunteered and consented to the study
* Measured at least 24 hours after antenatal corticosteroid and delivered within a maximum of 72 hours after measurement

Exclusion Criteria:

* Multiple pregnancies
* Amniotic fluid pathologies
* Fetal lung and liver diseases
* Fetal genetic and structural anomalies
* Signs and diagnoses of systemic maternal diseases
* Advanced maternal obesity preventing measurement
* Patients hospitalized with a diagnosis of preterm labor and discharged before delivery
* Presence of comorbid diseases of pregnancy (GDM, hypertensive diseases of pregnancy, PPROM, chorioamnionitis etc.)
* Pregnant women over 45 years of age, systemic conditions (history of chronic, mental, physical illness, severe renal, hepatic, gastrointestinal acute/chronic inflammatory disease, hyperthyroidism, hypothyroidism, hypertension, type 1/2 DM, history of malignancy, smoking, alcohol use)

Ages: 24 Weeks to 34 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will include single pregnant women with maternal age of 18-45 years, gestational age between 24-34 weeks, diagnosed with preterm labor, amniotic fluid pathology, fetal congenital and chromosomal anomalies, and fetuses without fetal congenital and chromosomal anomalies, who were hospitalized in the ward after the application to the Perinatology Clinic of Etlik City Hospital. A total of 80 patients without systemic maternal disease findings and diagnoses, without chronic drug use, who were measured at least 24 hours after antenatal corticosteroids were administered and delivered within a maximum of 72 hours, will be included in our study as two case groups with and without RDS diagnosis in neonatal follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-06 (Actual); Primary Completion 2024-03-06 (Estimated); Study Completion 2024-03-06 (Estimated)

PRIMARY OUTCOMES:
Fetal Lung Elastography Measurement | Prenatal (24-34 gestational weeks, before 72 hours to delivery)
  Measurement of prenatal ultrasonographic shear wave elastographic values(kPa) of the fetus in cases of preterm labor

CONTACTS AND LOCATIONS:
Overall Officials: Ahmet Kurt, 1, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Patient data is not open to sharing due to hospital policy. however, if necessary, the principal investigator can be reached via e-mail.